CLINICAL TRIAL: NCT03530761
Title: Kidney Biomarkers for the Prediction of Response to Terlipressin and Survival in Cirrhotic Patients With Acute Kidney Injury: Multicenter, Prospective Cohort Study
Brief Title: Korean Cohort Study of AKI & HRS in Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Sang Gyune Kim, Associate proffesor, Soonchunhyang University Hospital
Other Study IDs: P-KAKI
Record Dates: First submitted 2018-04-25; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Liver Cirrhosis; Acute Kidney Injury; Hepatorenal Syndrome
MeSH Terms: conditions — Liver Cirrhosis; Acute Kidney Injury; Hepatorenal Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute kidney injury: Increase in serum creatinine more than 0.3 mg/dl within 48 hours or a percentage increase serum creatinine more than 50% from baseline.
- Hepatorenal syndrome: 1. Diagnosis of cirrhosis and ascites,
  2. Diagnosis of AKI according to ICA-AKI criteria
  3. No response after 2 consecutive days of diuretic withdrawal and plasma volume expansion with albumin 1 g per kg of body weight
  4. Absence of shock
  5. No current or recent use of nephrotoxic drugs (non-steroidal anti-inflammatory drugs, aminoglycosides, iodinated contrast media, etc.)
  6. No macroscopic signs of structural kidney injury, defined as: absence of proteinuria (> 500 mg/day), absence of microhaematuria (> 50 RBCs per high power field), normal findings on renal ultrasonography.

SUMMARY:
The aim of this study is to investigate i) whether two biomarkers (urine NAG, urinary cystatin C) could be predictive factor in patient with liver cirrhosis, , and ii) whether these biomarkers can predict response of terlipressin.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) in patients with liver cirrhosis is sometimes accompanied by tubular injury which can lead to poor outcome. Current AKI criteria using serum creatinine (Cr) has some limitations to predict reversibility of renal function and discriminate renal parenchymal injury in cirrhotic patients. The aim of this study is to evaluate whether urine biomarkers [cystatin C, N-acetyl-β-D-Glucosaminidase (NAG)] can predict survival and response to terlipressin in cirrhotic patients with AKI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver cirrhosis diagnosed as acute kidney injury or hepatorenal syndrome
* Patients who voluntarily agreed to the study

Exclusion Criteria:

* Patients with active bleeding (eg, varix bleeding) within 7 days
* Patients with hepatocellular carcinoma
* Patients with hypersensitivity to terlipressin
* Patients with anuria
* Pregnant and lactating patients
* Patients who did not agree with the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis diagnosed as acute kidney injury or hepatorenal syndrome
Sampling Method: Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to 3 years
  From date of sample collection until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years

SECONDARY OUTCOMES:
Transplantation free survival | up to 3 years
  From date of sample collection until the date of first liver transplantation or date of death from any cause, whichever came first, assessed up to 3 years
Regression of acute kidney injury | up to 1 month
  Regression is defined as movement of AKI to a lower stage and decrease of serum creatinine
Recurrence of acute kidney injury | up to 1 year
  From sample collection day to elevation day of creatinine
Progression to chronic kidney disease | 1 year
  From sample collection day to progression to CKD
Response rate to terlipressin | 1 week
  If reduction of creatinine 0.3mg/dL from the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Ju Yoo, Doctor, Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- SoonChunHyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Helmersson-Karlqvist J, Arnlov J, Carlsson AC, Lind L, Larsson A. Urinary KIM-1, but not urinary cystatin C, should be corrected for urinary creatinine. Clin Biochem. 2016 Oct;49(15):1164-1166. doi: 10.1016/j.clinbiochem.2016.07.015. Epub 2016 Jul 28. PMID 27475248
- [Result] Ariza X, Sola E, Elia C, Barreto R, Moreira R, Morales-Ruiz M, Graupera I, Rodriguez E, Huelin P, Sole C, Fernandez J, Jimenez W, Arroyo V, Gines P. Analysis of a urinary biomarker panel for clinical outcomes assessment in cirrhosis. PLoS One. 2015 Jun 4;10(6):e0128145. doi: 10.1371/journal.pone.0128145. eCollection 2015. PMID 26042740
- [Result] Angeli P, Tonon M, Pilutti C, Morando F, Piano S. Sepsis-induced acute kidney injury in patients with cirrhosis. Hepatol Int. 2016 Jan;10(1):115-23. doi: 10.1007/s12072-015-9641-1. Epub 2015 Jul 4. PMID 26141259
- [Result] Wong F, Murray P. Kidney damage biomarkers: Novel tools for the diagnostic assessment of acute kidney injury in cirrhosis. Hepatology. 2014 Aug;60(2):455-7. doi: 10.1002/hep.27063. Epub 2014 Jun 18. No abstract available. PMID 24700173
- [Result] Wong F. The evolving concept of acute kidney injury in patients with cirrhosis. Nat Rev Gastroenterol Hepatol. 2015 Dec;12(12):711-9. doi: 10.1038/nrgastro.2015.174. Epub 2015 Oct 20. PMID 26484442
- [Result] Jaques DA, Spahr L, Berra G, Poffet V, Lescuyer P, Gerstel E, Garin N, Martin PY, Ponte B. Biomarkers for acute kidney injury in decompensated cirrhosis: A prospective study. Nephrology (Carlton). 2019 Feb;24(2):170-180. doi: 10.1111/nep.13226. PMID 29369449
- [Result] Belcher JM, Sanyal AJ, Peixoto AJ, Perazella MA, Lim J, Thiessen-Philbrook H, Ansari N, Coca SG, Garcia-Tsao G, Parikh CR; TRIBE-AKI Consortium. Kidney biomarkers and differential diagnosis of patients with cirrhosis and acute kidney injury. Hepatology. 2014 Aug;60(2):622-32. doi: 10.1002/hep.26980. Epub 2014 Jun 26. PMID 24375576
- [Result] Belcher JM, Garcia-Tsao G, Sanyal AJ, Thiessen-Philbrook H, Peixoto AJ, Perazella MA, Ansari N, Lim J, Coca SG, Parikh CR; TRIBE-AKI Consortium. Urinary biomarkers and progression of AKI in patients with cirrhosis. Clin J Am Soc Nephrol. 2014 Nov 7;9(11):1857-67. doi: 10.2215/CJN.09430913. Epub 2014 Sep 2. PMID 25183658
- [Result] Fagundes C, Pepin MN, Guevara M, Barreto R, Casals G, Sola E, Pereira G, Rodriguez E, Garcia E, Prado V, Poch E, Jimenez W, Fernandez J, Arroyo V, Gines P. Urinary neutrophil gelatinase-associated lipocalin as biomarker in the differential diagnosis of impairment of kidney function in cirrhosis. J Hepatol. 2012 Aug;57(2):267-73. doi: 10.1016/j.jhep.2012.03.015. Epub 2012 Apr 17. PMID 22521351
- [Result] Yap DY, Seto WK, Fung J, Chok SH, Chan SC, Chan GC, Yuen MF, Chan TM. Serum and urinary biomarkers that predict hepatorenal syndrome in patients with advanced cirrhosis. Dig Liver Dis. 2017 Feb;49(2):202-206. doi: 10.1016/j.dld.2016.11.001. Epub 2016 Nov 10. PMID 27876501
- [Result] Barreto R, Elia C, Sola E, Moreira R, Ariza X, Rodriguez E, Graupera I, Alfaro I, Morales-Ruiz M, Poch E, Guevara M, Fernandez J, Jimenez W, Arroyo V, Gines P. Urinary neutrophil gelatinase-associated lipocalin predicts kidney outcome and death in patients with cirrhosis and bacterial infections. J Hepatol. 2014 Jul;61(1):35-42. doi: 10.1016/j.jhep.2014.02.023. Epub 2014 Mar 5. PMID 24613364
- [Result] Angeli P, Gines P, Wong F, Bernardi M, Boyer TD, Gerbes A, Moreau R, Jalan R, Sarin SK, Piano S, Moore K, Lee SS, Durand F, Salerno F, Caraceni P, Kim WR, Arroyo V, Garcia-Tsao G. Diagnosis and management of acute kidney injury in patients with cirrhosis: revised consensus recommendations of the International Club of Ascites. J Hepatol. 2015 Apr;62(4):968-74. doi: 10.1016/j.jhep.2014.12.029. Epub 2015 Jan 28. No abstract available. PMID 25638527